CLINICAL TRIAL: NCT03964532
Title: TALAVE: A Pilot Trial of Induction Talazoparib Followed by Combination of Talazoparib and Avelumab in Advanced Breast Cancer
Brief Title: TALAVE: Induction Talazoparib Followed by Combination of Talazoparib and Avelumab in Advanced Breast Cancer
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Georgetown University (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00000023
Record Dates: First submitted 2019-04-22; First posted 2019-05-28 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Advanced Breast Cancer; Talazoparib; Avelumab
MeSH Terms: conditions — Breast Neoplasms | interventions — talazoparib; avelumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Phase I/Phase II (Experimental): Talazoparib (1mg by mouth [PO] daily D1-28) will be provided as monotherapy for the first cycle. Starting with cycle 2 and for all subsequent cycles, treatment with avelumab (800 mg intravenously [IV] D1 every 2 weeks) will be added to talazoparib.
  Interventions: Drug: Talazoparib; Drug: Avelumab

INTERVENTIONS:
Drug: Talazoparib — Talazoparib (formerly MDV3800 and BMN673) is an oral small molecule, selective inhibitor of PARP-1 and PARP-2.
  Other Names: Talzenna
Drug: Avelumab — Avelumab (formerly MSB0010718C) is a human immunoglobulin G1 (IgG1) anti-PD-L1 monoclonal antibody131 that utilizes both adaptive and innate immune mechanisms.
  Other Names: Bavencio

SUMMARY:
This is a multi-institutional pilot trial for patients with advanced breast cancer. The trial is designed to assess the safety and tolerability of induction talazoparib followed by combination of talazoparib and avelumab. As an exploratory endpoint, the study team will evaluate the immunomodulatory effects of induction talazoparib followed by the combination of talazoparib and avelumab in patients with advanced breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed advanced breast cancer not amenable to curative treatment by surgery or radiotherapy, that is amenable to biopsy
* Radiographically measurable disease by RECIST v1.1
* Age ≥ 18 years
* Life expectancy of more than 3 months
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 1
* Signed informed consent form
* Patients with a standard 12-lead electrocardiogram (ECG) with the following parameters at screening (defined as the mean of the triplicate ECGs):

  1. QTc interval at screening < 481 msec
  2. Resting heart rate 50-100bpm
* Adequate hepatic, bone marrow, and renal function at the time of enrollment:

  1. Bone Marrow: Absolute neutrophil count (ANC) ≥ 1,500/mm3; Platelets ≥ 100,000/mm3; Hemoglobin ≥ 9.0 g/dL. Patients must be able to meet the criteria without transfusion or receipt of colony stimulating factors within 2 weeks before obtaining sample
  2. Creatinine clearance ≥ 60 mL/min based on Cockcroft-Gault equation
  3. Hepatic function: aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 × the upper normal limit of institution's normal range. Total bilirubin ≤ 1.5 × the upper normal limit of institution's normal range, except for subjects with documented history of Gilbert's syndrome who may enroll at Investigator discretion. For subjects with liver metastases, AST and ALT < 5 × the upper normal limit of institution's normal range, and total bilirubin >1.5 - 3.0 x the upper normal limit of institution's normal range are acceptable as long as there is no persistent nausea, vomiting, right upper quadrant pain or tenderness, fever, rash, or eosinophilia
  4. Prothrombin Time (PT) and Partial Thromboplastin Time (PTT) must be ≤ 2 X the upper limit of the institution's normal range and International Normalized Ratio (INR) < 2. Subjects on anticoagulation (such as coumadin) will be permitted to enroll as long as the INR is in the acceptable therapeutic range as determined by the investigator
* Patients may have received an unlimited number of prior therapies. The last dose of systemic therapy must have occurred a minimum of 2 weeks prior to C1D1.
* Patients must have fully recovered from all effects of surgery. Patients must have had at least two weeks after minor surgery and four weeks after major surgery before starting therapy. Minor procedures requiring conscious sedation such as endoscopies or mediport placement may only require a 24-hour waiting period, but this must be discussed with an investigator
* Women of childbearing potential must have a negative serum pregnancy test within 14 days prior to initiation of treatment and/or postmenopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential
* Patient is capable of swallowing pills whole
* Subject, or legally authorized representative (LAR) is capable of understanding and complying with parameters as outlined in the protocol and able to sign and date the informed consent, approved by the IRB, prior to the initiation of any screening or study-specific procedures
* Patient, or LAR, must consent to multiple biopsies during study.

Exclusion Criteria:

* Prior disease progression while receiving anti-PD-1 or anti-PD-L1 therapy within 6 months of use
* Prior exposure to PARP inhibitor-based therapy
* Patients with known untreated central nervous system (CNS) metastases
* Recent severe infection or antibiotic use, or known chronic infection with human immunodeficiency virus (HIV) or hepatitis B virus
* Signs or symptoms of infection within 2 weeks prior to Cycle 1, Day 1
* Diagnosis of immunodeficiency or is receiving systemic steroid or other immunosuppressive therapy
* Active autoimmune disease that has required systemic treatment in the past 2 years
* History of tuberculosis
* History of allogenic bone marrow transplant or solid organ transplant
* History of idiopathic pulmonary fibrosis, pneumonitis (including drug induced), organizing pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia, etc.), or evidence of active pneumonitis on screening chest CT scan
* Life-threatening visceral disease or other severe concurrent disease that would, in the investigator's judgment, cause unacceptable safety risks, contraindicate patient participation in the clinical study or compromise compliance with the protocol
* Live vaccine administration within 30 days of planned start of study therapy
* Cardiovascular disease problems including unstable angina, therapy for lifethreatening ventricular arrhythmia, or myocardial infarction, stroke within the last 6 months, or a diagnosis of congestive heart failure
* Patient has impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of the study drugs
* Presence of a psychiatric illness or social situation that would limit compliance with study requirements
* Women who are pregnant or breastfeeding
* Patients with history of another active malignancy within the past 2 years, excluding non-melanoma carcinoma of the skin
* Patients receiving any other investigational agents
* Patients must not have had radiotherapy encompassing >20% of the bone marrow
* Patients must not have current evidence of any condition, therapy, or laboratory abnormality (including active or uncontrolled myelosuppression [ie, anemia, leukopenia, neutropenia, thrombocytopenia]) that might confound the results of the study or interfere with the patient's participation for the full duration of the study treatment or that makes it not in the best interest of the patient to participate
* Patients must not be considered a poor medical risk due to a serious, uncontrolled medical disorder, nonmalignant systemic disease, or active, uncontrolled infection.
* Current use of potent P-gp inhibitors within 7 days prior to randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-04-17 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Quantification of Grade 3 and 4 toxicities (Adverse Events) | from the start of study drugs through 30 days after end of treatment (approximately 1 year)
  Quantification of grade 3 and 4 toxicities according to the National Cancer Institute Common Toxicity Criteria for Adverse Events Version 4.0 [NCI CTCAE v4.03]. Toxicity analysis will be conducted in all patients receiving at least one dose of talazoparib.

SECONDARY OUTCOMES:
The anti-tumor efficacy as measured by Objective Response Rate (ORR). | 4 Months
  Objective response rate (ORR) at 4 months, defined as the proportion of patients with a documented PR or CR according to the RECIST version 1.1 and irRECIST; as a total cohort and BRCA1/2 carriers versus wildtype.

OTHER OUTCOMES:
The anti-tumor efficacy as measured by Progression Free Survival (PFS). | Up to 5 years
  Progression free survival (PFS) is defined as the time from cycle 1 day 1 to determination of tumor progression by RECIST version 1.1 or death due to any cause, whichever occurs first
The anti-tumor efficacy as measured by Overall Survival (OS). | Up to 5 years
  Overall survival. OS is defined by time from study enrollment till death from any cause
The anti-tumor efficacy as measured by Duration of Response (DOR). | Up to 5 years
  Duration of response (DOR) by RECIST is defined as the time from first documentation of CR or PR by RECIST v1.1 until the time of first documentation of disease progression per RECIST v1.1
The anti-tumor efficacy as measured by Disease Control Rate (DCR). | 4 months
  Disease control rate (DCR) is defined as the proportion of patients with a documented CR, PR, or SD at 4 months according to the RECIST version 1.1 and irRECIST

CONTACTS AND LOCATIONS:
Overall Officials: Claudine Isaacs, MD, Principal Investigator — Georgetown University
Locations (2):
- United States (2):
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - University of Utah, Huntsman Cancer Institute, Salt Lake City, Utah